CLINICAL TRIAL: NCT05615194
Title: A Randomized Clinical Study to Assess the Impact of a Single Dexmedetomidine Bolus During Induction of General Anesthesia on Intraoperative Sevoflurane Consumption in Elective Laparoscopic Surgery
Brief Title: The Impact of a Single Dexmedetomidine Bolus on Intraoperative Sevoflurane Consumption (DEXHALE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Olivier Verdonck, Assistant Professor, Deputy chief of the Department of Anesthesiology of Maisonneuve-Rosemont Hospital, University of Montreal(UDeM), Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-3190
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Inhalation Anesthesia; Dexmedetomidine; Sevoflurane; Laparoscopy
Keywords: Environment; kgCO2eq
MeSH Terms: interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be 1:1 randomly assign to one of the two following groups: dexmedetomidine 0.6 mcg.kg-1 (group D) or a saline placebo of equivalent volume (group C) to be administered on 10 minutes during induction.
  The patient presenting all the inclusion criteria and no exclusion criteria for this study will be approached by the anesthesia research team. They will provide explanations on the study as well as a consent form to the patient for him to have time to read it before the surgery. The risk of serious and unexpected adverse reactions to dexmedetomidine will also be disclosed to the patient before his agreement to participate to the study. After his approval, the patient will sign the consent and will be randomized.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient, the anesthesiologist in charge, the surgeon, the PACU staff and the research team evaluating the patient in PACU will be blinded to the randomization group.
  The syringe containing the dexmedetomidine or the placebo will be prepared by an anesthesiologist or a pharmacist external to the study and identified by a unique number so that the patient's group can be identified if needed. Both solutions are translucent and total volume to be administered on 10 minutes during induction will be of equal volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline in volume equivalent of dexmedetomidine dose according to patient weight ; Administered via infusion pump (Smith Medical Medfusion® 4000 Syringe Infusion Pump) so that the full dose is delivered over 10 minutes during induction of general anesthesia
  Interventions: Drug: Placebo
- Dexmedetomidine (Active Comparator): Dexmedetomidine 0.6 mcg/kg (adjusted body weight) ; Administered via infusion pump (Smith Medical Medfusion® 4000 Syringe Infusion Pump) so that the full dose is delivered over 10 minutes during induction of general anesthesia
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 0.6 mcg/kg in infusion over 10 minutes
  Other Names: Precedex; Dexmedetomidine Hydrochloride; DIN : 02339366
  Arms: Dexmedetomidine
Drug: Placebo — Volume equivalent in infusion over 10 minutes
  Other Names: Normal Saline; NaCl 0.9%
  Arms: Placebo

SUMMARY:
Sevoflurane is a volatile agent easy to control thanks to the Minimum Alveolar Concentration (MAC) allowing its titration for an optimal depth of anesthesia. Growing biomedical evidence also highlight its anti-inflammatory and antioxidant effects protecting against ischemia-reperfusion injury in cardiac surgery and, potentially, in organ transplant. The estimated annual contribution of inhalational anesthetic agents represents about 0.01% of global CO2 production. Alternatives such as total intravenous anesthesia (TIVA) avoid direct greenhouse emission, but their indirect carbon footprint remains a major problem. For all these reasons, this research aim to find a way to maintain the use of sevoflurane for its clinical benefits while reducing its consumption to limit the environmental consequences. The use of dexmedetomidine could help anesthesiologists to achieve this greener sevoflurane anesthesia. Dexmedetomidine is a potent, highly selective α-2 adrenergic receptor agonist described as a unique sedative with analgesic and sympatholytic properties. This new randomized controlled trial (RCT) will answer the question whether a single bolus of dexmedetomidine (0.6 mcg.kg-1 on 10 minutes during induction) compared to placebo has a clinically significant impact on sevoflurane consumption during laparoscopic elective surgery.

DETAILED DESCRIPTION:
Inhaled gases have been used since the advent of anesthesia due to their analgesic and dissociative properties. However, these are now part of a growing environmental debate which leads us to reconsider their systematic use for general anesthesia. Sevoflurane is a volatile agent easy to monitor using the Minimal Alveolar Concentration (MAC) facilitating its titration for adequate anesthesia depth. Growing biomedical evidence also highlight its anti-inflammatory and antioxidant effects protecting against ischemia-reperfusion injury in cardiac surgery and, potentially, in organ transplant.

The estimated annual contribution of inhalational anesthetic agents represents about 0.01% of global CO2 production. This data can be illustrated as a commercial airliner flying 418 times around the world. Desflurane is gradually abandoned as its greenhouse effect is 25 times more potent than sevoflurane for an equivalent MAC and fresh gas flow. As low-flow inhalational techniques and scavenging technologies become the standard of practice, anesthesiologists still cannot prevent the gas to be released in the atmosphere .

Alternatives such as total intravenous anesthesia (TIVA) avoid direct greenhouse emission, but their indirect carbon footprint remains a major problem. Propofol has a high potential for bioaccumulation. It has high mobility in soil, resists degradation in aquatic environment and concentrates in adipose tissue of aquatic organism. To control its toxicity, destruction should be done by incineration over 1000°C. Unfortunately, studies prove that 32-49% of dispensed propofol is waisted and is mostly disposed unproperly.

For all these reasons, this research aim to find a way to maintain the use of sevoflurane for its clinical benefits while reducing its consumption to limit the environmental consequences.

The use of dexmedetomidine could help us achieve this greener sevoflurane anesthesia. Dexmedetomidine is a potent, highly selective α-2 adrenergic receptor agonist described as a unique sedative with analgesic and sympatholytic properties. Currently approved for sedation, this molecule shows many advantages compared to hypnotic drugs such as propofol. Although still under investigation, dexmedetomidine would possibly have a lower hazard environmental score. The use of dexmedetomidine also shows promising results regarding the reduction of emergence cough and agitation. Decrease in pain and post-operative nausea and vomiting (PONV) are other benefits of dexmedetomidine providing conditions to promote enhanced recovery after surgery (ERAS).

Many investigations have studied impacts of dexmedetomidine as an adjuvant to general anesthesia for its opioid sparing capacity, and hemodynamics response during laparoscopic surgeries. Fewer research specifically wondered about sevoflurane dispense outcome. Moreover, they don't reflect the anesthesia practice of North America and their sample sizes are low.

This new randomized controlled trial (RCT) will answer the question whether a single bolus of dexmedetomidine (0.6 mcg.kg-1 on 10 minutes during induction) compared to placebo has a clinically significant impact on sevoflurane consumption during laparoscopic elective surgery. Opioid requirement, need for vasopressors, post-operative events (PONV, shivering, critical respiratory event) and time for readiness for Post-Anesthesia Care Unit (PACU) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients
* Undergoing laparoscopic surgery of duration time expected under 120 minutes using general anesthesia with sevoflurane
* Fully consented
* Age > 18yo
* No allergy to one of the medications used in this study.

Exclusion Criteria:

* History of severe coronary artery disease; ventricular dysfunction, serious cardiac arrhythmia (including atrial fibrillation and high-grade atrioventricular block)
* Moderate to severe renal or hepatic dysfunction
* Allergy to any drug used in the study protocol
* Refusal of the patient for participation in the study
* History of severe PONV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Sevoflurane consumption expressed in mL.kg-1.h-1 | From intubation to end of surgery
  To compare the total sevoflurane consumption when using a dexmedetomidine single bolus (group D) of 0.6 mcg.kg-1 on 10 minutes during induction versus placebo (group C). This will be expressed in mL.kg-1.h-1 of surgery.

SECONDARY OUTCOMES:
Total intra-operative remifentanil consumption (in mcg.kg-1) | From intubation to end of surgery
  To compare the total intra-operative remifentanil consumption during anesthesia based on the NoL index (Medasense Ltd., Ramat Gan, Israel)
Percentage of time during the intraoperative period for which the NOL index will be above the pain threshold of 25 (in % of surgical time) | From intubation to end of surgery
  To compare the percentage of time during the intraoperative period for which the NOL index will be above the pain threshold of 25
Total amount of hydromorphone given IV in PACU (in mg) | From PACU admission to discharge
  To quantify the total amount of hydromorphone needed in PACU
Intra-operative and postanesthesia care unit (PACU) doses of vasopressors | From intubation to PACU discharge
  To compare the intra- and post-operative requirements of phenylephrine, ephedrine, glycopyrrolate and atropine
Mean end tidal sevoflurane (in %) and MAC needed to maintain the BIS index (Medtronic, Canada) between 40 and 60 | From intubation to end of surgery
  To compare the mean end tidal sevoflurane (EtSevo) and MAC needed to maintain the BIS index between 40 and 60
Total intraoperative time from intubation until end of surgery with BIS index between 40 and 60 (in minutes) | From intubation to end of surgery
  To compare the % of total intraoperative time from intubation until end of surgery with BIS index between 40 and 60
Time for extubation (in minutes) | From sevoflurane discontinuation to extubation
  To compare the time for extubation
Time for awakening (in minutes) | From sevoflurane discontinuation to when the patient is opening his eyes
  To compare the time for awakening
Postoperative outcomes such as postoperative nausea and vomiting (PONV), shivering and critical respiratory event (CRE) | From PACU admission to discharge
  To assess postoperative outcomes such as postoperative nausea and vomiting (PONV), shivering and critical respiratory event (CRE)
  A CRE will be defined as the occurrence of one of the following criteria:
  * Upper airway obstruction requiring an intervention
  * Moderate hypoxemia: SpO2 of 90-93% on 2 L.min-1 nasal cannula O2
  * Severe hypoxemia: SpO2 < 90% on 2 L.min-1 nasal cannula O2
  * Signs of respiratory distress or impeding ventilatory failure
  * Patient requiring reintubation in the PACU
  * Clinical evidence or suspicion of pulmonary aspiration after tracheal extubation
Total time spent in PACU (in minutes) | From PACU admission to discharge
  To compare total time for readiness for discharge from PACU between groups assessed by recovery scores (Aldrete's modified score and Maisonneuve-Rosemont PACU score)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Maisonneuve-Rosemont, CIUSSS de l'Est de l'Ile de Montréal, Montreal, Quebec, Canada